CLINICAL TRIAL: NCT05937425
Title: The Effect of Nurse Navigation Program Applied in Line With Supportive Care Needs in Patients Diagnosed With Lung Cancer on Anxiety-Depression, Adaptation to the Disease and Quality of Life
Brief Title: The Effect of Nurse Navigation Program on Lung Cancer Patients
Acronym: [LungCaNN]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Müge ALTINIŞIK, MSc, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 240778
Record Dates: First submitted 2023-06-22; First posted 2023-07-10 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Cancer; Nurse Navigator; Nurse Navigation Program; Individualized Care; Anxiety-Depression; Adaptation to the Disease; Quality of Life
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial consisting of two groups: experimental and control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Effects of nurse navigation program on patients with lung cancer
  Interventions: Other: LungCaNN
- Control group (No Intervention): An information note will be given to the control group.

INTERVENTIONS:
Other: LungCaNN — The needs of the patients included in the study will be determined with the supportive care needs scale. A training booklet will be given to the patients in the intervention group and they will be informed about the existing or newly formed unsupported care needs, the evaluation of their frequency and severity, and the ability of the patients to call the navigator nurse 24/7 or send an SMS. For interventions that can be applied in line with evidence-based guidelines for unsupported care needs with patients included in the intervention group every week for 12 weeks, a face-to-face navigation will be made by the navigator nurse over the phone and once a month.
  Arms: Intervention group

SUMMARY:
The study aims to determine the effect of the nurse navigation program (LungCaNN), which is performed in line with the supportive care needs of newly diagnosed non-small cell lung cancer patients, on the level of anxiety-depression, adherence to the disease, and quality of life.

The study was designed as a randomized study with a control group. This study will be carried out with a total of 84 NSCLC patients, 42 of whom were in the intervention group and 42 in the control group, whose treatment was started in Akdeniz University Medical Oncology Outpatient Clinic and met the inclusion criteria of the sampling. Nurse navigation program will be applied for 12 weeks from the diagnosis of NSCLC patients in the intervention group. The intervention protocol of the study is abbreviated as "Lung Cancer Nurse Navigator" [LungCaNN].

Within the scope of the LungCaNN program, face-to-face patient education, patient education booklet, face-to-face, and telephone navigation initiatives were planned. Patient Identification Form, Depression Anxiety Stress Scale (DASS 21), Chronic Disease Adjustment Scale, EORTC QLQ 30 Quality of Life Scale-/ LC-13, and Navigation and Interview Steps Form will be used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Know how to read and write No hearing or speech problems Be able to use the phone The primary medical diagnosis is non-small cell lung cancer Karnofsky Performance Scale score of 70% or higher Patients with a stress thermometer of 4 and above At most six weeks past the date of diagnosis

Exclusion Criteria:

* Patients with cognitive problems Expected life expectancy is less than three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Depression, Stress, Anxiety Scale (DASS21) | change from baseline DASS21 at 12 week
  It is used to evaluate depression, stress, and anxiety levels. Each item scores between 0-3 and gives separate scores for depression, stress, and anxiety. A maximum of 21 and a minimum of 0 points can be obtained from the scales. High scores indicate high levels of depression, stress, and anxiety.
EORTC QLQ - C30 Quality of Life Scale/ LC-13 Lung Module | change from baseline EORTC QLQ - C30 Quality of Life Scale/ LC-13 Lung Module at 12 week
  This scale was developed to measure the quality of life of cancer patients. It includes 30 questions and three sub-dimensions: General Well-being, Functional Difficulties, and Symptom Control. The maximum score on the scale is 100 and the minimum score is 0. High scores in the functional subscale indicate good/healthy functional status, high scores in the symptom subscale indicate high levels of symptoms and/or problems, and high scores in the global health status/quality of life subscale indicate good quality of life. Scoring of the Quality of Life Scale LC-13 Lung Module is also done by symptom scale scoring. A high score from the LC-13 Lung Module indicates that the symptoms are experienced intensely.
Scale of Adjustment to Chronic Diseases | change from baseline Scale of Adjustment to Chronic Diseases at 12 week
  The scale was developed to determine the level of compliance of patients with the disease. It consists of 25 items. It consists of three sub-dimensions: Physical Adaptation, Social Adaptation, and Psychological Adaptation. The total score that can be obtained from the scale is 125. High scores from the sub-dimensions and/or the whole scale mean that the patient's level of compliance with the disease also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Arikan, PhD, RN, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Konyaalti, Antalya, Turkey (Türkiye)